CLINICAL TRIAL: NCT03761927
Title: Effect of Noise Reduction Algorithms on Physiological, Behavioural and Subjective Measures of Listening Effort
Brief Title: Physiological, Behavioural and Subjective Measures of Listening Effort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Sonova2018_36
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hearing Aid without NR enabled. (Active Comparator): Hearing Aid without Noise Reduction (NR) enabled serves as reference condition.
  Interventions: Device: Hearing Aid without NR enabled
- Hearing Aid with NR(1) (Experimental): Hearing Aid with Noise Reduction I (NR) enabled.
  Interventions: Device: Hearing Aid with NR(1)
- Hearing Aid with NR(2) (Experimental): Hearing Aid with Noise Reduction II (NR) enabled.
  Interventions: Device: Hearing Aid with NR(2)

INTERVENTIONS:
Device: Hearing Aid without NR enabled — Each participant will be fitted with noise reduction disabled. Disabled means that no sound processing algorithm that removes noise from the speech signal is active.
  Arms: Hearing Aid without NR enabled.
Device: Hearing Aid with NR(1) — Each participant will be fitted with the noise reduction program on the same hearing aid. The principle of the noise reduction algorithm is to remove noise from a speech signal with the aim of improving the speech intelligibility and comfort.
  Arms: Hearing Aid with NR(1)
Device: Hearing Aid with NR(2) — Each participant will be fitted with a second noise reduction program on the same hearing aid. The parameterization of this NR algorithm differs from that in NR(1).
  Arms: Hearing Aid with NR(2)

SUMMARY:
Participants will perform two different listening tasks: (1) listening to, and repeating back, sentence lists presented in noise, and (2) listening to short radio excerpts and answering subsequent comprehension questions. At the same time participants are required to perform a manual target-tracking task on a touch screen. During this study, continuous, non-invasive physiological measurements (heart rate, skin conductance and hemoencephalography) will be made from participants. Using this paradigm we will be assessing the effect of different hearing aid processing algorithms on listening effort. The study takes the form of a three factor (listening task x algorithm x signal-to-noise ratio), within-subjects design. Each participant performs each listening task (about 4min long each) with each algorithm (reference, noise reduction I, noise reduction II), at two signal-to-noise ratios (+4 decibel and 0 decibel) twice (test-retest).

ELIGIBILITY:
Inclusion Criteria:

* Healthy outer ear (without previous surgical procedures)
* Ability to fill in a questionnaire conscientiously
* Informed Consent as documented by signature
* Minimum 1 year hearing aid experience
* Moderate-Severe (N3-N5) hearing loss or Normal Hearing

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments
* Inability to produce a reliable hearing test result
* Massively limited dexterity
* Known psychological problems
* Known central hearing disorders

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Heart rate variability data | 6 weeks
  Heart rate variability will be recorded from the participant both before and during the performance of the auditory tasks. Analyses will be carried out relative to the baseline recording (made before the auditory tasks), in order to account for differences in baseline physiological activity. Heart rate variability will be analysed in both the time [ms] and frequency [ms squared] domains.
Skin conductance data | 6 weeks
  Skin conductance will be recorded from the participant both before and during the performance of the auditory tasks. Analyses will be carried out relative to the baseline recording (made before the auditory tasks), in order to account for differences in baseline physiological activity. It is planned to analyse mean levels of skin conductance [micro-Siemens].

SECONDARY OUTCOMES:
Hemoencephalography data | 6 weeks
  Hemoencephalography will be recorded from the participant both before and during the performance of the auditory tasks. Analyses will be carried out relative to the baseline recording (made before the auditory tasks), in order to account for differences in baseline physiological activity. Hemoencephalography will be analysed simply as the ratio of the blue and red light [%] during auditory task performance.
Dual-task performance test 1 | 6 weeks
  Performance on the secondary tracking task will be analysed in order to observe whether there is a dual-task cost associated with performing both tasks simultaneously. Typically the level of degradation on the secondary task is thought to reflect an increased listening effort (provided that the primary task performance remains stable). Accordingly, success on the primary task will also be monitored and used in analyses (speech intelligibility in [%] correct). For the Secondary task performance the reaction time [ms] will be analysed.
Dual-task performance test 2 | 6 weeks
  Performance on the secondary tracking task will be analysed in order to observe whether there is a dual-task cost associated with performing both tasks simultaneously. Typically the level of degradation on the secondary task is thought to reflect an increased listening effort (provided that the primary task performance remains stable). Accordingly, success on the primary task will also be monitored and used in analyses (comprehension questions [numbers] correct after listening to radio excerpts). For the Secondary task performance the reaction time [ms] will be analysed.
Subjective Listening Effort rating | 6 weeks
  Subjective Listening Effort will also be assessed through self-reported individual listening effort on a 14 point scale from "only noise" to "no effort" after each auditory task.

CONTACTS AND LOCATIONS:
Overall Officials: Juliane Raether, Principal Investigator — Sonova AG
Locations (1):
- Sonova AG, Stäfa, Switzerland

IPD SHARING:
Plan to Share IPD: No